CLINICAL TRIAL: NCT07358208
Title: Prospective Familial Cohort for Pancreas Research
Brief Title: Prospective Familial Registry for Pancreas Research
Acronym: PARTNER
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-002416
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Family History of Pancreas Cancer
Keywords: Family history of pancreas cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — One-time specimen up to 50cc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family history of pancreas cancer: Prospective cohort of individuals who do not have pancreas cancer but are members of a kindred with two or more blood-related family members with pancreas cancer, or with at least one blood-related family member with pancreas cancer and one relative who carries a variant in a gene known to be associated with pancreatic cancer.

SUMMARY:
The purpose of this research is to develop a resource registry of individuals currently without pancreatic cancer but are members of a kindred with two or more blood-related family members with pancreas cancer.

DETAILED DESCRIPTION:
If you agree to be in the study, you will be asked to fill out a questionnaire once every two years. The questionnaire will ask you questions about your health and family history. The investigator may ask you to donate a one-time blood specimen of approximately 3½ tablespoons, which can be done at your local doctor's office. The investigator may ask you if you are willing to provide the names and addresses of other family members who may be eligible to participate in the study. No visits to Mayo Clinic are required for your participation.

ELIGIBILITY:
Inclusion Criteria:

1. An individual who was previously enrolled in Mayo Clinic IRB # 1197-00, 354-06, 355-06, or 19-010791
2. Is age 18 years or older.
3. Has a valid United States mailing address.
4. Has at least two blood-related relatives who have had pancreas cancer or has a blood-relative with pancreatic cancer and that relative carries a known germline mutation in APC, ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2, PMS2, STK11, TP53 or mutations in other genes known to be associated with pancreatic cancer.

Exclusion Criteria:

1. An individual who is a prison inmate
2. An individual who is not compos mentis (of sound mind, memory, and understanding), and not able to give consent.
3. Has personal history of pancreas cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US citizens who meet eligibility requirements
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2040-11 (Estimated); Study Completion 2040-11 (Estimated)

PRIMARY OUTCOMES:
To establish a prospective cohort of individuals from pancreas cancer families | 25 years
  To establish and actively follow a resource registry of individuals currently without pancreatic cancer but are members of a kindred with two or more blood-related family members with pancreas cancer.
Change in health | 25 years
  Participants will be asked to complete a health questionnaire every 2 years to ascertain new cancer diagnosis in the subject and in first-degree relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Antwi, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials